CLINICAL TRIAL: NCT03648138
Title: Testing the Influence of Different Sugary Drink Warning Label Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Drexel University (Other); New York University (Other); University of Connecticut (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christina Roberto, Assistant Professor of Medical Ethics and Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 828087; R01DK111558 (NIH)
Record Dates: First submitted 2018-08-07; First posted 2018-08-27 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Weight Gain; Diabetes Type 2
MeSH Terms: conditions — Obesity; Weight Gain; Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: Although participants are not blinded to the study arm to which they are randomized, they are not told the true purpose of the study until after completing the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie label (Active Comparator): This arm will display a "Calories per Bottle" label on all beverages, not just sugary beverages. This label is identical to the American Beverage Association's current "Clear on Calories" labels (as of 2018).
  Interventions: Behavioral: Sugary drink warning labels
- Text warning label (Experimental): This arm will display similar text proposed in a recent sugary drink warning label bill in California. Sample text: WARNING: Drinking beverages with added sugar(s) contributes to obesity, type 2 diabetes, and tooth decay. The calorie label will also appear on all beverages.
  Interventions: Behavioral: Sugary drink warning labels
- Sugar graphic warning label (Experimental): This arm will graphically display the amount of sugar in each sugary beverage along with the same text used in the "text warning label" arm. The calorie label will also appear on all beverages.
  Interventions: Behavioral: Sugary drink warning labels
- Health graphic warning label (Experimental): This arm will graphically display potential negative health effects of over consuming sugary drinks for each sugary beverage, along with the same text used in the "text warning label" arm. The calorie label will also appear on all beverages.
  Interventions: Behavioral: Sugary drink warning labels

INTERVENTIONS:
Behavioral: Sugary drink warning labels — This information appears in the description of the study arms.

SUMMARY:
The aim of this study is to compare different sugary drink labels to see which most influence knowledge, beliefs, purchase intentions and choices. Parents of children ages 6-11 will shop in a virtual convenience store after being randomized to 1 of 4 conditions: 1) calorie labels; 2) text warning labels; 3) graphic sugar warning labels; or 4) graphic health warning. This study will provide data comparing the influence of sugary drink text warning labels and two kinds of graphic warning labels.

ELIGIBILITY:
Inclusion Criteria:

1. a primary caregiver of a child 6-to-11 years old;
2. ≥18 years old; and
3. can read and speak English

Exclusion Criteria:

1. not a primary caregiver of a child 6-to-11 years old;
2. <18 years old; and
3. cannot read and/or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Hypothetical beverage choice | The survey will take up to 20 minutes
  Participants will select a beverage to purchase in the virtual store. Our outcome will be the percentage of parents choosing a 20-ounce sugary drink for their child

SECONDARY OUTCOMES:
Likely to serve or buy these beverages: | The survey will take up to 20 minutes
  Item: "How likely are you to serve or buy this product for your child in the next 4 weeks?" This will be answered on a 7-point Likert scale.
Parent feels good serving the beverages | The survey will take up to 20 minutes
  Item: "Serving this product to my child would make me feel like I am doing something good for my child." This will be measured on a 7-point likert scale.
Child enjoyment of beverages | The survey will take up to 20 minutes
  Item: "How much do you think your child would enjoy this product?" This will be answered on a 7-point likert scale.
Health beliefs and risk perceptions index | The survey will take up to 20 minutes
  We will create this outcome by summing responses to the following 7 health perception questions 6 prompted with the statement "Drinking this product often would…". The statements end with the following health belief and risk perception language: "lead my child to gain weight," "increase my child's risk of heart disease," "increase my child's risk of diabetes," "make my child feel energized," "help my child focus at school", and "help my child live a healthy life." The other item is: "How healthy do you think this product is for your child?" Responses to questions about weight gain, heart disease, and diabetes will be reverse coded, so higher scores on the index will indicate a stronger positive health perception of the beverages. These will be scored on 7-point likert scales.
Estimate of how many teaspoons of added sugar are in the beverages | The survey will take up to 20 minutes
  This variable will be measured continuously based on a text box provided to participants.
Perceived amount of added sugar in beverages | The survey will take up to 20 minutes
  This variable will be measured on a 3-point Likert scale ranging from "too little for my child" to "too much for my child".
Noticing the label | The survey will take up to 20 minutes
  Participants will respond "yes," "no," or "I don't know" to the item: "When you selected a beverage to buy for your child at the beginning of this survey, did you notice any labels on the beverages other than calorie information?"
Perceived label influence | The survey will take up to 20 minutes
  Participants will respond: "yes", "no," or "I did not notice any labels" in response to the question of whether the label influenced their purchase.
Favor or oppose sugary drink warning label policy | The survey will take up to 20 minutes
  We will compare the percentage of participants in favor of (combining somewhat favor and strongly favor), opposed to (combining somewhat oppose and strongly oppose), or neutral about the policy based on the following question: "Would you favor or oppose a government policy requiring a warning label to be placed on beverages with added sugars?" Ratings will be from -2 to 2.
Likelihood of label changing thoughts | The survey will take up to 20 minutes
  Item: "If this government warning label were on a beverage, how much would it change your thoughts about the healthiness of that beverage for your child?" This will be measured on a 5-point Likert scale.
Encourage you to give fewer beverages to your child | The survey will take up to 20 minutes
  Item: "If you saw this government warning label on a beverage, would the label encourage you to serve your child that beverage less often?" The responses will be measured on a 5-point Likert scale.
How much do you trust the information on this label | The survey will take up to 20 minutes
  Item: "How much do you trust the information on this label?". Responses will be measured on a 7-point Likert scale.
Negative reactions to the label | The survey will take up to 20 minutes
  We will examine the average negative emotional response to the label (said the warning label made them feel worried, fearful, guilty, or disgusted or grossed out). Each emotion will be scored on a 5-pt likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Online study with GfK, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified dataset via an online data storage website (e.g., open science framework, dataverse, research box)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available soon after the paper is published in a peer-reviewed journal.
Access Criteria: All researchers will be able to access the data.

REFERENCES:
- [Derived] Musicus AA, Gibson LA, Bellamy SL, Orr JA, Hammond D, Glanz K, Volpp KG, Schwartz MB, Bleakley A, Strasser AA, Roberto CA. Effects of Sugary Beverage Text and Pictorial Warnings: A Randomized Trial. Am J Prev Med. 2023 May;64(5):716-727. doi: 10.1016/j.amepre.2023.01.018. Epub 2023 Feb 8. PMID 36764835